CLINICAL TRIAL: NCT04140045
Title: The Effect of Hypohydration During Cycling in the Heat on Acute Kidney Injury Biomarkers
Brief Title: The Effect of Manipulating Hydration Status During Cycling in the Heat on Acute Kidney Injury Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Loris Juett, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R19-P130
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Hypohydrated; Euhydrated
MeSH Terms: interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypohydrated (Experimental): Participants will be required to restrict their water intake during cycling in the heat (90-120 minutes at 35°C), in order to achieve a body mass loss of approximately 3%.
  Interventions: Other: Water intake
- Euhydrated (Experimental): Participants will be provided with water intake that matches their sweat losses during cycling in the heat (90-120 minutes at 35°C)
  Interventions: Other: Water intake

INTERVENTIONS:
Other: Water intake — Water intake will be manipulated in both arms to create a hypohydrated state and a euhydrated state, post-exercise

SUMMARY:
Acute Kidney Injury (AKI) is common in prolonged endurance events. Risk factors for exercise-associated AKI include: the exercise itself, heat, hypohydration, muscle breakdown and non-steroidal anti-inflammatory drug (NSAID) use. Prior research from our laboratory showed the hypohydration during high-intensity running increased a biomarker of AKI (urine osmolality-corrected kidney injury molecule 1). Therefore, the current study will now investigate the effect of manipulating hydration status during cycling on biomarkers of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* recreationally active

Exclusion Criteria:

* Smoker/vaper
* regular use of anti-inflammatory medications (e.g. ibuprofen)
* history of kidney disease or diabetes

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Changes in urinary Kidney Injury Molecule 1 (uKIM-1) (uncorrected/raw values and urine osmolality-corrected values) | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
  A novel protein biomarker for acute kidney injury
Changes in urinary neutrophil gelatinase-associated lipocalin (uNGAL) (uncorrected/raw values and urine osmolality-corrected values) | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
  A novel protein biomarker for acute kidney injury
Changes in urine osmolality | Pre-exercise (baseline) and post-exercise (immediately after the intervention), as well as all urine produced from post-exercise until 24 hours post-baseline
  A measure of urine concentration.
Changes in serum creatinine | Pre-exercise (baseline), post-exercise (immediately post-exercise), 24 hours post-baseline
  Serum creatinine is a marker of kidney function
Incidence of Acute Kidney Injury (as determined by changes in serum creatinine) | Pre-exercise (baseline), post-exercise (immediately post-exercise), 24 hours post-baseline
  A rise in serum creatinine of 1.5 fold or more from baseline will be defined as acute kidney injury

SECONDARY OUTCOMES:
Plasma volume changes | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
Changes in serum osmolality | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
  The gold standard marker of hydration status
Body mass changes | pre-exercise (baseline), throughout exercise, post-exercise (immediately after the intervention), 24 hours post-baseline
Changes in creatine kinase | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
  A marker of muscle damage
Changes in lactate dehydrogenase | Pre-exercise (baseline), post-exercise (immediately after the intervention), 24 hours post-baseline
  A marker of muscle damage
Ad libitum energy (Kj), carbohydrate (g), sugar (g), protein (g), fat (g), saturated fat (g), sodium (g) and water intake (g). | from post-exercise (immediately after the intervention) until 24 hours post-baseline
  Participants will complete a weighed food and fluid diary, using a set of food scales and a diary, to record all food and fluid that they ingest. This data will then be analysed using dietary analysis software (e.g. Nutritics)
Changes in headache scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their headache on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in nausea scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their nausea on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in dizziness scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their dizziness on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in thirst scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their thirst on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in thermal comfort scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their thermal comfort on a scale of -10 to 10, with -10 being cold impossible to bear and 10 being heat impossible to bear
Changes in gastrointestinal comfort scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their gastrointestinal comfort on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in stomach fullness scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their stomach fullness on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in stomach bloatedness scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their stomach bloatedness on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in urge to vomit scores | pre-exercise (baseline), every 30 minutes during exercise (30, 60,90 and 120 minutes), post-exercise (immediately after the intervention) and 24 hours post-baseline
  Participants will be asked to rate their urge to vomit on a scale of 0-10, with higher scores meaning a worse outcome .
Changes in urinary creatinine | pre-exercise (baseline), post-exercise (immediately after the intervention) and 24 hours post-baseline
Changes in heart rate | Will be monitored throughout the exercise intervention, at 15 minute intervals (15 minutes, 30 minutes, 45 minutes, 60 minutes, 75 minutes, 90 minutes, 105 minutes and 120 minutes)
  Provides insight into exercise intensity
changes in rating of perceived exertion | Will be monitored throughout the exercise intervention, at 30 minute intervals (30 minutes, 60 minutes, 90 minutes and 120 minutes)
  Provides insight into exercise intensity
Changes in aural temperature | Will be determined immediately prior to the exercise intervention (at rest) and then throughout the exercise intervention at 15 minute intervals (15 minutes, 30 minutes, 45 minutes, 60 minutes, 75 minutes, 90 minutes, 105 minutes and 120 minutes)
  in-ear temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, United Kingdom